CLINICAL TRIAL: NCT00137397
Title: A Multi-centre, Randomised, Placebo Controlled, Double Blind, Parallel Group Study in Female Patients to Evaluate Whether Tolterodine ER Can Reverse the Increased Bladder Wall Thickness in Patients With Overactive Bladder.
Brief Title: A Study to Measure the Effect of Tolterodine Extended Release on the Thickness of the Bladder Wall in Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121006
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Tolterodine ER
Drug: Placebo

SUMMARY:
The main aim of the study is to investigate whether taking Tolterodine for overactive bladder symptoms can reduce the thickness of the bladder wall, as measured by intra-vaginal ultrasound. This will help doctors to understand whether there is a link between changes in the thickness of the bladder wall and progression of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder (described as urinary urgency, with or without urge incontinence, usually with frequency and nocturia for more than 6 months
* Bladder wall thickness of 5mm or more

Exclusion Criteria:

* Treatment in the previous four weeks with an anticholinergic drug or any drug for the treatment of overactive bladder.
* Significant stress incontinence - Urinary tract infection or a history of intermittent urinary tract infections (more than four episodes in the last two years).
* Conditions considered significant by the investigator (e.g. cystocoele, significant bladder prolapse, bladder stone, indwelling catheter etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-11; Study Completion 2006-08

PRIMARY OUTCOMES:
The main outcome will be the change in bladder wall thickness, as measured by intra-vaginal ultrasound from baseline to week 12.

SECONDARY OUTCOMES:
Secondary outcomes are the change in bladder wall thickness, as measured by intra-vaginal ultrasound from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United Kingdom (10):
  - Pfizer Investigational Site, Blackburn, Lancashire
  - Pfizer Investigational Site, Harrow, Middx
  - Pfizer Investigational Site, Oxford, Oxfordshire
  - Pfizer Investigational Site, Livingston, West Lothian
  - Pfizer Investigational Site, Basingstoke
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Cambs
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Northampton
  - Pfizer Investigational Site, Pl6 8Dh

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121006&StudyName=A+study+to+measure+the+effect+of+Tolterodine+ER+on+the+thickness+of+the+bladder+wall+in+patients+with+overactive+bladder